CLINICAL TRIAL: NCT05847868
Title: Clinical Evaluation of Moment Tumor Hip Replacement Products Within the Scope of Substantial Clinical Trials
Brief Title: Clinical Evaluation of Moment Tumor Hip Replacement Products
Acronym: KRIOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Estas Tıbbi Mamülleri Medikal (Industry)
Collaborators: Klinar CRO (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: K-BE001-KRIOS
Record Dates: First submitted 2023-04-07; First posted 2023-05-08 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Primary and Secondary Bone Tumor in the Proximal Femur Region
Keywords: hip; pain; fracture; inability; proximal
MeSH Terms: conditions — Pain; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Device Feasibility (Experimental): Device feasibility will be performed in this single arm study.
  Interventions: Device: Moment Tumour Hip Prothesis

INTERVENTIONS:
Device: Moment Tumour Hip Prothesis — In the case of irreversible bone loss due to bone tumors, large and multi-part fractures, and pseudarthrosis in the proximal region of the femur bone, the defective bone area is removed and implants made of artificial materials are placed in order to replace the integrity of the bone. In addition, implant applications are made to the proximal femur region for the purpose of revision arthroplasty, which is typically replaced by total hip prosthesis depending on the wear condition.
  In this way, the bone integrity will be preserved, long-term stabilization will be provided to the patient and existing pain will be eliminated.
  Moment Tumor Hip Replacement Systems consist of proximal main body, extension pieces and intramedullary stems. Components are available in a variety of sizes to meet anatomical requirements and surgeon needs.

SUMMARY:
The aim is to ensure that the patients are functionally adequately and painlessly mobilized with the proximal femoral tumor resection prosthesis used, to increase the survival of patients who underwent wide resection, and to determine the complications of the treatment applied and the clinical performance of the Moment Tumor Hip Replacement Products used.

DETAILED DESCRIPTION:
This study is a 6-center, prospective local medical device clinical trial. Trial period is 6 months. Patient recruitment will continue until the target sample number determined by the power analysis is reached. Since the application is surgical, it is within the scope of a one-time application. The patients will be followed for 6 months from the day of surgery. The study was designed as a prospective cohort study planned to be cross-sectional. The aim of this study is to ensure that the patients are functionally adequately and painlessly mobilized with the proximal femoral tumor resection prosthesis used, to increase the survival of patients who underwent wide resection, and to determine the complications of the treatment applied and the clinical performance of the Moment Tumor Hip Replacement Products used and to contribute to the medical literature on proximal femoral resection prosthesis as a result of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults of both sexes aged 18-79 years
* For patients with bone loss, fractures, pseudarthrosis due to primary-secondary metastases in the hip femoral region, patients belonging to one or more of the following groups
* Patients with or with bone resections due to infection
* Patients with unsuccessful femoral component applications
* Patients in need of long-term stabilization of major bone defects caused by fractures with major and irreversible bone loss, periprosthetic fractures, traumatic non-tumor conditions affecting the trunks of the long bones, and comminuted fractures
* Patients with severe pain and loss of function in the proximal femoral region
* Patients with incompetence of the upper end of the femur or femoral neck fracture in hip replacement revisions.
* Have sufficient mental and physical capacity to sign the informed consent form for the procedure

Exclusion Criteria:

* Be under the age of 18 and over the age of 79
* Pregnancy
* Breastfeeding
* Patients with bone tumors near the implant
* Patients with acute or chronic infections (local or systemic) that reduce the adhesion resistance of the implant.
* Patients with defective bone structures that may prevent proper fixation of the implant and severe deterioration or axial deviation affecting bone quality
* Patients with inadequate bone quantity and quality as a result of osteoporosis
* Patients with underdeveloped skeletal structure
* Patients with vascular and neuromuscular disorders or muscular dystrophy and advanced muscle atrophy
* Patients with impaired blood flow caused by vascular changes due to previous surgical procedure, alcohol use, etc.
* Patients with more than expected implant overload due to obesity and/or vigorous physical activity or strain (such as sports, activities requiring physical activity)
* Patients with inflammatory degenerative joint disease
* Patients with pathologies that prevent surgical intervention
* Patients whose general condition is not good and who cannot handle anesthesia
* Patients who are uncoordinated or unwilling to operate, or who cannot follow instructions
* Patients with mental retardation who do not or cannot comply with post-operative care instructions
* Patients with neuropathic osteoarthropathy (charcot joint) joint disease
* Patients with multiple organ failure
* Patients with sepsis
* Patients with syndromes or concomitant diseases that may adversely affect the evaluation of patients due to its systematic involvement.
* Patients whose follow-up is not clinically or ethically appropriate due to complications that may develop during the study

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of Adverse Events | 6 Months
  Reliability of the procedure (adverse events occurring)
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 6 Months
  Toleratibily of the patients for the procedure.
Hip pain and function for 6 months after the procedure according to the MSTS scoring | 6 Months
  Hip pain and function for 6 months after the procedure according to the MSTS scoring
Change in Quality of life | 6 Months
  Determination of the change in quality of life from baseline to 6 month after the procedure

SECONDARY OUTCOMES:
Improvement in Functional Parameters | 6 Months
  Percent change in in functional parameters compared to baseline during the follow-up period.
Complications | 6 Months
  Complications will be evaluated in patients with complications according to the Henderson classification.
Procedure's Safety | 6 Months
  Number of adverse event: observed adverse events (AE) with the help of radiographic evaluations and Examinations performed

CONTACTS AND LOCATIONS:
Locations (7):
- Turkey (Türkiye) (7):
  - Gazi University Faculty of Medicine, Ankara
  - Hacettepe University Faculty of Medicine, Ankara
  - Pamukkale University Faculty of Medicine, Denizli
  - Eskişehir Osmangazi University Health Practice and Research Hospital, Eskişehir
  - Istanbul Göztepe Prof.Dr. Suleyman Yalcin City Hospital, Istanbul
  - Necmettin Erbakan University Meram Faculty of Medicine, Konya
  - Cumhuriyet University School of Medicine, Sivas

IPD SHARING:
Plan to Share IPD: No
There i no plan to share IPD